CLINICAL TRIAL: NCT03368677
Title: Targeting SPMS: Effect of Teriflunomide Treatment on Microglial Activation in an MS Patient Cohort at Risk of Progression. A [11C]PK11195 Brain PET Study
Brief Title: Effect of Teriflunomide Treatment on Microglial Activation in an MS Patient Cohort at Risk of Progression
Acronym: TERIPET
Status: Active, not recruiting | Type: Observational
Sponsor: Turku University Hospital (Other Government)
Responsible Party: Sponsor
Other Study IDs: TERIPET
Record Dates: First submitted 2017-10-02; First posted 2017-12-11 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-04

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood, urine and faecal samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Teriflunomide group: 20 MS patients who are using teriflunomide medication under the supervision of their treating neurologist.
- No disease modifying treatment: 10 MS-patients who do not use any regular disease modifying MS treatment of their own volition

SUMMARY:
To evaluate the effect of teriflunomide treatment on microglial activation in late stage multiple sclerosis.

DETAILED DESCRIPTION:
In Multiple Sclerosis (MS), plaques in the white and grey matter of the brain represent the best known pathological changes of the disease, but a significant inflammation process has also been detected outside these plaques in connection with the disease. This extensive, diffuse inflammatory process correlates with the progression of the disease, measured by EDSS score (Expanded Disability Status Scale status) and reduction in patients' cognitive level. According to neuropathological research, the diffuse inflammatory process outside the plaques is connected with powerful activation of microglia, oxidative stress, and deficiencies in mitochondrial activity. The activation of microglial cells can be measured in vivo in patients using positron-emission tomography (PET) scanning and so-called TSPO radioligands, such as the 11C-PK11195 radioligand. 11C-PK11195 radioligand binds to TSPO molecules, which manifest on the surface of activated, but not un-activated, microglia.

Teriflunomide treatment is expected to slow down the process of increasing microglial activation. TSPO-PET imaging allows in vivo follow-up of the pathogenic process associated with the gradual MS disease evolution, and allows to evaluate whether teriflunomide treatment has an effect on disease progression-related pathology.

ELIGIBILITY:
Inclusion Criteria:

* Signing the consent form
* Having used teriflunomide treatment for at least 6 months
* 40-55 years of age at the time of signing the research consent form
* MS diagnosis in accordance with either the Poser or McDonald criteria
* EDSS 2-6.5
* Clear lesion load in brain MRI (> 9 T2 lesion)

Exclusion Criteria:

* Patients suffering from another brain disease of in addition to multiple sclerosis
* Steroid treatment 4 weeks prior to the scan
* Significant pathology in the MRI scan other than MS-related lesions
* Patients suffering from claustrophobia or panic disorder, or patients who have exhibited hypersensitivity of PET markers (practical obstacle to the scan)
* Exposure to experimental radioactivity in the last 12 months such that the dosimetry threshold would be exceeded due to participation in the study
* Severe hepatic impairment
* Pregnant women, or women of childbearing potential who are not using reliable contraception during treatment with teriflunomide and thereafter as long as its plasma levels are above 0.02 mg/l.

Ages: 40 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The research will recruit MS patients who are using teriflunomide treatment and are followed-up at the Neurology Outpatient Clinic at the Turku University Hospital. The study will not interfere with the initiation or dosage of the medication in any manner. The patient's treating neurologist will select the most suitable medication on the basis of the patient's clinical status, and patients using teriflunomide medication will be offered the option to participate in this imaging research.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2017-12-01 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Change of 11C-PK11195-radioligand binding using PET | 0 to 12 months
  Change in microglia-activity in late RRMS patients on teriflunomide treatment during one-year interval as measured by PET imaging and [11C]PK11195 radioligand.

SECONDARY OUTCOMES:
MRI metrics | 0, 12 months, 24 months, 36 months
  To evaluate lesion load of the white matter MS plaques
EDSS | 0, 12 months, 24 months, 36 months
  Expanded Disability Status Scale
BICAMS | 0, 36 months
  Brief International Cognitive Assessment for MS

CONTACTS AND LOCATIONS:
Overall Officials: Laura Airas, MD,professor, Principal Investigator — Turku University Hospital, division of clinical neurosciences
Locations (1):
- Turku PET Centre, Turku, Southwest Finland, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Sjoros T, Saraste M, Matilainen M, Nylund M, Koivumaki M, Kuhle J, Leppert D, Airas L. Serum glial fibrillary acid protein associates with TSPO-expressing lesions in multiple sclerosis brain. Ther Adv Neurol Disord. 2025 Jul 28;18:17562864251352998. doi: 10.1177/17562864251352998. eCollection 2025. PMID 40756531